CLINICAL TRIAL: NCT05966480
Title: A Phase 2, Multicenter, Multinational, Randomized, Double-blind, Placebo-Controlled Study to Assess the Safety, Efficacy, and Pharmacokinetics of Multiple Dose Levels of ESK-001 in Adult Patients With Systemic Lupus Erythematosus
Brief Title: Phase 2 Placebo-Controlled Study to Assess the Safety and Efficacy of ESK-001 in Active Systemic Lupus Erythematosus
Acronym: LUMUS
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Alumis Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ESK-001-010
Record Dates: First submitted 2023-06-29; First posted 2023-07-28 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: SLE
Keywords: Autoimmune Diseases; Immune System Diseases; Connective Tissue Diseases; Immune-mediated Diseases; Active Systemic Lupus Erythematosus; SLE; Lupus; LUMUS; Lupus Erythematosus, Systemic
MeSH Terms: conditions — Autoimmune Diseases; Immune System Diseases; Connective Tissue Diseases; Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- ESK-001 Dose Level 1 (Experimental): ESK-001 administered as an oral tablet
  Interventions: Drug: ESK-001
- ESK-001 Dose Level 2 (Experimental): ESK-001 administered as an oral tablet
  Interventions: Drug: ESK-001
- ESK-001 Dose Level 3 (Experimental): ESK-001 administered as an oral tablet
  Interventions: Drug: ESK-001
- Placebo (Placebo Comparator): Placebo administered as an oral tablet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ESK-001 — Oral tablet
  Arms: ESK-001 Dose Level 1; ESK-001 Dose Level 2; ESK-001 Dose Level 3
Drug: Placebo — Oral tablet
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the clinical efficacy, safety, PK, and PD of multiple dose levels of ESK-001 compared with placebo in adult patients with SLE.

DETAILED DESCRIPTION:
This study will consist of a 5 week screening period, 48 week treatment period, and a 4 week follow up period for a total of 57 weeks. Each participant will be randomized to receive ESK-001 or placebo for 48 weeks. An open label extension study will be available for those patients who complete the study.

ELIGIBILITY:
Inclusion Criteria:

Patients with 6 or more months of SLE according to the 2019 EULAR/ACR criteria, have positive autoantibodies or low complement at screening, and have active SLE as measured by SLEDAI-2K of 6 or more, or 4 or more if joint involvement is present.

Patients need to be on treatment which can be:

* A stable dose of oral corticosteroid (≤40 mg/day prednisone or equivalent) for a minimum of 2 weeks prior to signing of the informed consent form (ICF) at the Screening Visit. The dose of oral corticosteroid the patient is taking should not increase between screening and Week 0 (Day 1).
* And/or antimalarial treatment (e.g., hydroxychloroquine, chloroquine, quinacrine),
* And/or no more than 1 of the following conventional DMARDS:

  * Azathioprine ≤200 mg/day
  * Mycophenolate mofetil ≤2 g/day or mycophenolic acid ≤1.44 g/day
  * Oral, subcutaneous, or intramuscular (IM) methotrexate ≤20 mg/week.

Exclusion Criteria:

* Drug-induced SLE or other autoimmune diseases that, in the opinion of the Investigator, are likely to confound efficacy assessments
* Active, proliferative lupus nephritis that in the Investigator's opinion may require treatment not allowed by the protocol
* Current disease other than SLE that, in the opinion of the Investigator, is likely to interfere with SLE disease activity assessments. Examples include severe fibromyalgia, severe osteoarthritis and severe cardiorespiratory diseases.
* Active severe or unstable neuropsychiatric SLE including, but not limited to the following: aseptic meningitis; cerebral vasculitis; myelopathy; demyelination syndromes (ascending or transverse myelitis, acute inflammatory demyelinating polyradiculopathy); acute confusional state; impaired level of consciousness; psychosis; acute stroke or stroke syndrome; cranial neuropathy; new seizures; cerebellar ataxia; and mononeuritis multiplex.

  * That would make the patient unable to fully understand the ICF, or
  * Where, in the opinion of the Principal Investigator, protocol-specified SOC is insufficient and utilization of a more aggressive therapeutic approach not permitted in the protocol, is indicated
* Known history of a primary immunodeficiency or an underlying condition such as HIV infection or splenectomy that predisposes the patient to infection
* Currently active, clinically significant infection of any kind
* Clinically significant chronic infection (eg, osteomyelitis, bronchiectasis) within 8 weeks prior to signing the ICF (chronic fungal nail infections are allowed)
* Any infection requiring hospitalization or treatment with IV anti-infectives not completed at least 4 weeks prior to signing the ICF
* Any infection requiring oral anti-infectives (including antivirals) within 2 weeks prior to Day 1
* Any severe herpes infection at any time prior to Week 0 (Day 1), including, but not limited to, disseminated herpes (ever), herpes encephalitis (ever), recurrent herpes zoster (defined as 2 episodes within 2 years), or ophthalmic herpes (ever)

  * Active herpes zoster infection within 12 weeks of prior to signing the ICF
  * Active herpes simplex virus within 4 weeks of Day 1
* Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408 (Actual)
Dates: Start 2023-06-26 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
To compare the effect on disease activity measured by the proportion of patients achieving British Isles Lupus Assessment Group (BILAG)-based Composite Lupus Assessment (BICLA) response at Week 48 between doses of ESK-001 and placebo | Week 48

SECONDARY OUTCOMES:
To assess the safety and tolerability of multiple dose levels of ESK-001 | Week 48
  Safety and Tolerability will be assessed with clinical and laboratory assessments including blood tests for liver and kidney function, ECGs, hematological measures and physical examinations throughout the time of the study and safety follow up. The number and proportion of TEAEs, SAEs, AEs of greater than grade 3 severity and AEs of Clinical Interest will be recorded.
To compare the effect on disease activity measured by the proportion of patients achieving an SLE Responder Index of ≥4 (SRI[4]) response at Week 48 | Week 48
To compare corticosteroid use in patients at Week 48 | Week 48
  To compare the number and percentage of patients using corticosteroids and continuous summaries of dose used will be assessed as well as the frequency and percentage of patients able to taper corticosteroids and maintain low doses following taper.
To compare the effect on cutaneous disease activity measured by the proportion of patients with a CLASI activity score of ≥8 at baseline achieving ≥ 50% reduction in the CLASI activity score at Week 48 between doses of ESK-001 and placebo | Week 48
To compare the effect on disease activity measured by the proportion of patients achieving BICLA responses at Week 48 between doses of ESK-001 and placebo by stratification groups | Week 48
To compare the Lupus Low Disease Activity State (LLDAS) response between doses of ESK-001 and placebo at Week 48 | Week 48
To compare the annualized flare rate through Week 48 | Week 48
To use the SF-36 (Short Form-36 item QoL measure) to compare the effect on health-related quality of life (HRQOL) between doses of ESK-001 and placebo | Week 48
  Efficacy: Comparing the effects of Esk-001 doses vs Placebo on Patient Reported Outcome (PRO) as it relates to Health-Related Quality of Life (HRQoL) as measured by self-reporting using the SF-36 (Short Form-36 item QoL measure) Questionnaire which uses a scale of 0 to 100. The higher numbers mean better health.
To use the SLE-specific Lupus Quality of Life (LQoL) questionnaire to compare the effect on health-related quality of life (HRQOL) between doses of ESK-001 and placebo | Week 48
  Efficacy: Comparing the effects of Esk-001 doses vs Placebo on Patient Reported Outcome (PRO) as it relates to Health-Related Quality of Life (HRQoL) as measured by self-reporting using the SLE-specific Lupus Quality of Life (LQoL) questionnaire which uses a scale of 0 to 100. The higher numbers mean better health.
To compare disease-specific QoL between doses of ESK-001 and placebo | Week 48
  Efficacy: To compare disease-specific QoL between doses of ESK-001 and placebo using the SLE Disease Activity Index 2000 (SLEDAI2K) measured on a scale of 0 to 105 where the higher numbers mean more disease activity.
To compare disease-specific QoL between doses of ESK-001 and placebo | Week 48
  Efficacy: To compare disease-specific QoL between doses of ESK-001 and placebo using the British Isle Lupus Assessment Group 2004 (BILAG-2004) with a scale of A to E (A meaning very active disease and E no current or previous disease).
To compare disease-specific QoL between doses of ESK-001 and placebo | Week 48
  Efficacy: To compare disease-specific QoL between doses of ESK-001 and placebo using the Physician's Global Assessment (PGA) evaluating disease response using the 4-point VAS (Visual Analog Scale) of 0 to 3 (0 means no flares and 3 means severe flare in disease).
To compare Fatigue measured by FACIT-F between doses of ESK-001 and placebo | Week 48
  To compare patient-reported fatigue as measured by Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) questionnaire between doses of ESK-001 and placebo, where the score range is 0 to 52 and a lower score indicates greater fatigue/worse outcome.
To compare patient global assessment of disease activity (PtGA) between doses of ESK-001 and placebo | Week 48
  Efficacy: To compare disease-specific QoL between doses of ESK-001 and placebo using the PtGA (Patient Global Assessment) instrument. Patients record on a visual analog scale (VAS) how well or badly they feel as a result of the disease in their own estimation over the course of the study.

CONTACTS AND LOCATIONS:
Locations (169):
- United States (48):
  - Investigator Site #1046, Anniston, Alabama
  - Investigator Site #1104, La Jolla, California
  - Investigator Site #1050, Los Alamitos, California
  - Investigator Site #1168, Mission Hills, California
  - Investigator Site #1174, Napa, California
  - Investigator Site #1061, Upland, California
  - Investigator Site #1048, Aventura, Florida
  - Investigator Site #1063, Avon Park, Florida
  - Investigator Site #1176, Bradenton, Florida
  - Investigator Site #1045, Clearwater, Florida
  - Investigator Site #1055, Coral Gables, Florida
  - Investigator Site #1097, Coral Springs, Florida
  - Investigator Site #1091, Daytona Beach, Florida
  - Investigator Site #1051, DeBary, Florida
  - Investigator Site #1087, Hollywood, Florida
  - Investigator Site #1135, Kissimmee, Florida
  - Investigator Site #1060, Miami, Florida
  - Investigator Site #1093, Miami, Florida
  - Investigator Site #1057, Miami, Florida
  - Investigator Site #1067, Miami Lakes, Florida
  - Investigator Site #1090, Plantation, Florida
  - Investigator Site #1089, Tampa, Florida
  - Investigator Site #1170, Atlanta, Georgia
  - Investigator Site #1052, College Park, Georgia
  - Investigator Site #1204, Chesterfield, Missouri
  - Investigator site #1209, Las Vegas, Nevada
  - Investigator Site #1189, Sparta, New Jersey
  - Investigator Site #1101, Albuquerque, New Mexico
  - Investigator Site #1058, Brooklyn, New York
  - Investigator Site #1088, New York, New York
  - Investigator Site #1175, Queens, New York
  - Investigator Site #1095, Charlotte, North Carolina
  - Investigator Site #1056, Charlotte, North Carolina
  - Investigator Site #1173, Charlotte, North Carolina
  - Investigator Site #1171, Philadelphia, Pennsylvania
  - Investigator Site #1062, Pittsburgh, Pennsylvania
  - Investigator Site #1044, Memphis, Tennessee
  - Investigator Site #1195, Carrollton, Texas
  - Investigator Site #1049, Colleyville, Texas
  - Investigator Site #1071, Fort Worth, Texas
  - Investigator Site #1094, Houston, Texas
  - Investigator Site #1169, Houston, Texas
  - Investigator site #1178, Houston, Texas
  - Investigator Site #1187, Red Oak, Texas
  - Investigator site #1053, San Antonio, Texas
  - Investigator Site #1186, San Antonio, Texas
  - Investigator Site #1172, Spring, Texas
  - Investigator Site #1194, Tomball, Texas
- Argentina (8):
  - Investigator Site #3012, CABA, Buenos Aires
  - Investigator Site #3001, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Investigator Site #3016, La Plata, Buenos Aires
  - Investigator Site #3009, San Miguel de Tucumán, Tucman
  - Investigator Site #3010, San Miguel de Tucumán, Tucman
  - Investigator Site #3015, San Miguel de Tucumán, Tucumán Province
  - Investigator Site #3023, Buenos Aires
  - Investigator Site #3008, Mendoza
- Bulgaria (7):
  - Investigator Site #5603, Haskovo
  - Investigator Site #5602, Pleven
  - Investigator Site #5525, Plovdiv
  - Investigator Site #5521, Plovdiv
  - Investigator Site #5529, Rousse
  - Investigator Site #5522, Sofia
  - Investigator Site #5547, Sofia
- Chile (2):
  - Investigator Site #3006, Providencia
  - Investigator Site #3002, Santiago
- Colombia (7):
  - Investigator Site #3019, Barranquilla
  - Investigator Site #3011, Barranquilla
  - Investigator Site #3021, Bogotá
  - Investigator Site #3022, Bogotá
  - Investigator Site #3020, Cali
  - Investigator Site #3003, Chía
  - Investigator Site #3014, Medellín
- Croatia (2):
  - Investigator Site #5542, Rijeka
  - Investigator Site #5543, Split
- Denmark (2):
  - Investigator Site #4012, Aarhus
  - Investigator Site #4011, Køge
- Georgia (6):
  - Investigator Site #5516, Tbilisi
  - Investigator Site #5523, Tbilisi
  - Investigator Site #5538, Tbilisi
  - Investigator Site #5536, Tbilisi
  - Investigator Site #5534, Tbilisi
  - Investigator Site #5517, Tbilisi
- Germany (3):
  - Investigator Site #4003, Leipzig
  - Investigator Site #4005, Mainz
  - Investigator Site #4006, Munich
- Hungary (2):
  - Investigator Site #5548, Debrecen
  - Investigator Site #5544, Gyula
- India (16):
  - Investigator Site # 6015, New Delhi, National Capital Territory of Delhi
  - Investigator Site #6005, Ahmedabad
  - Investigator Site #6010, Ahmedabad
  - Investigator Site #6016, Ahmedabad
  - Investigator Site #6006, Ahmedabad
  - Investigator Site #6001, Bangalore
  - Investigator Site #6009, Bengaluru
  - Investigator Site #6012, Chandigarh
  - Investigator Site #6004, Haryāna
  - Investigator Site #6013, Jaipur
  - Investigator Site #6011, Lucknow
  - Investigator Site #6008, Nagpur
  - Investigator Site #6014, Pune
  - Investigator Site #6007, Pune
  - Investigator Site #6002, Surat
  - Investigator Site #6003, Surat
- Mexico (16):
  - Investigator Site #2501, Chihuahua City
  - Investigator Site #2504, Cuauhtémoc
  - Investigator Site #2502, Guadalajara
  - Investigator Site #2512, Guadalajara
  - Investigator Site #2507, Guadalajara
  - Investigator Site #2508, Madero
  - Investigator Site #2509, Mexico City
  - Investigator Site #2514, Mexico City
  - Investigator Site #2503, Mexico City
  - Investigator Site #2506, Mexico City
  - Investigator Site #2511, Mérida
  - Investigator Site #2516, Mérida
  - Investigator Site # 2517, Naucalpan
  - Investigator Site #2510, Oaxaca City
  - Investigator Site #2505, San Luis Potosí City
  - Investigator Site #2513, Torreón
- Peru (5):
  - Investigator Site #3013, Lima
  - Investigator Site #3004, Lima
  - Investigator Site #3018, San Martín de Porres
  - Investigator Site #3005, Santiago de Surco
  - Investigator Site #3017, Trujillo
- Philippines (7):
  - Investigator Site #8003, Angeles City
  - Investigator Site #8009, Iloilo City
  - Investigator Site #8011, Lipa City
  - Investigator Site #8001, Manila
  - Investigator Site #8010, Manila
  - Investigator Site #8018, Manila
  - Investigator Site #8006, Quezon City
- Poland (14):
  - Investigator Site #5519, Bialystok
  - Investigator Site #5546, Bialystok
  - Investigator Site #5518, Bialystok
  - Investigator Site #5531, Bydgoszcz
  - Investigator Site #5520, Bytom
  - Investigator Site #5539, Częstochowa
  - Investigator Site #5533, Krakow
  - Investigator Site #5537, Nadarzyn
  - Investigator Site #5545, Poznan
  - Investigator Site #5535, Sosnowiec
  - Investigator Site #5532, Szczecin
  - Investigator Site #5527, Warsaw
  - Investigator Site #5540, Warsaw
  - Investigator Site #5528, Wroclaw
- Puerto Rico (2):
  - Investigator site #3028, Caguas
  - Investigator site #3029, San Juan
- Romania (3):
  - Investigator Site #5530, Bucharest
  - Investigator Site #5549, Bucharest
  - Investigator Site #5526, Bucharest
- South Korea (5):
  - Investigator Site #8007, Anyang-si
  - Investigator Site #8004, Busan
  - Investigator Site #8016, Seoul
  - Investigator Site #8019, Seoul
  - Investigator Site #8012, Seoul
- Spain (5):
  - Investigator Site #4013, A Coruña
  - Investigator Site #4008, Alicante
  - Investigator Site #4007, Barcelona
  - Investigator Site #4002, Seville
  - Investigator Site #4009, Valencia
- Taiwan (5):
  - Investigator Site #8013, Chiayi City
  - Investigator Site #8014, Kaohsiung City
  - Investigator Site #8008, Taichung
  - Investigator Site #8015, Taichung
  - Investigator Site #8017, Taipei
- United Kingdom (4):
  - Investigator Site #4017, Leeds
  - Investigator Site #4015, London
  - Investigator Site #4016, London
  - Investigator Site #4014, Southampton

IPD SHARING:
Plan to Share IPD: No